CLINICAL TRIAL: NCT04012866
Title: Effects of the Combined Cognitive Training and Aerobic Exercise on Cognition, Physiological Markers, Daily Function, and Quality of Life in Stroke Patients With Mild Cognitive Impairment
Brief Title: Effects of Combined Cognitive Training With Aerobic Exercise in Stroke Patients With MCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 107044-F
Record Dates: First submitted 2019-05-20; First posted 2019-07-09 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-06

CONDITIONS: Stroke
Keywords: Cognitive Rehabilitation; Aerobic Exercise; Computerized Cognitive Training
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SEQ (sequential training group) (Experimental): The sequential training group (SEQ) will first receive 30-minutes aerobic exercise training followed by 30-minutes computerized cognitive training. All participants will receive a training session for 60 minutes per day, two or three days per week for 12-18 weeks, a total of 36 training sessions.
  Interventions: Behavioral: Aerobic exercise training; Behavioral: Computerized cognitive training
- DUAL (dual training group) (Experimental): The dual training group (DUAL) will receive aerobic exercise training and computerized cognitive training simultaneously. All participants will receive a training session for 60 minutes per day, two or three days per week for 12-18 weeks, a total of 36 training sessions.
  Interventions: Behavioral: Aerobic exercise training; Behavioral: Computerized cognitive training
- CI (control intervention group) (Active Comparator): The control intervention group (CI) will receive a control training session for 60 minutes per day, two or three days per week for 12-18 weeks, a total of 36 training sessions.
  Interventions: Behavioral: Control training

INTERVENTIONS:
Behavioral: Aerobic exercise training — The aerobic exercise program using progressive resistive stationary bicycle training which will contain warm-up, resistive physical exercise, and cool-down. The training resistance will increase with improvement of participants' performance.
  Arms: DUAL (dual training group); SEQ (sequential training group)
Behavioral: Computerized cognitive training — The computerized cognitive training program will be implemented with the brainHQ to target abilities of visuospatial processing, attention, memory, and executive function. The level of the training program will become more difficult with progress in participants' targeted cognitive abilities.
  Arms: DUAL (dual training group); SEQ (sequential training group)
Behavioral: Control training — The Control training will receive an intervention including combinations of non-aerobic physical activities and unstructured mental activities.
  Arms: CI (control intervention group)

SUMMARY:
Cognitive impairments have severe impact on functional recovery and quality of life after stroke. Current evidence indicated that combining exercise and cognitive training may provide additional benefits on cognition in stroke. This study aims to investigate the effects and mechanisms of two combined methods of computer-based cognitive training with physical exercise in stroke patients with cognitive impairments.

DETAILED DESCRIPTION:
Cognitive impairment is not uncommon after stroke. Stroke patients with cognitive decline may experience difficulties in learning motor tasks, functional disability, and poor quality of life. Interventions for cognitive impairment remain under development and pharmaceutical intervention is not yet optimal at present. Targeted cognitive treatments or aerobic exercise training provided potential benefits to enhance cognitive function for stroke patients with cognitive decline. Recent studies demonstrate that combining exercise and cognitive training may provide additional benefits on cognition than single type of training. However, physical exercise training and cognitive-based intervention can be combined either sequentially or simultaneously. It remains unclear whether the two combination methods induce similar or differential effects in brain plasticity, physiological modulation, and behavioral outcomes for individuals with stroke. It is important to examine the potential effects, comparative effects and the neural mechanism of two combined interventions that can possibly maximize benefits for stroke survivors with cognitive impairments.

The purposes of the present study are to: (1) examine and compare the effects of two combined interventions on brain plasticity, physiological biomarkers and behavioral outcomes, including cognitive, physical, and daily functions, and quality of life, from pre- to post-training; (2) understand the neural mechanisms of cognitive recovery following two combined interventions using the electroencephalography (EEG); (3) examine the long-term benefits following the two combined interventions; (4) to identify the correlations between brain activity, biomarkers and behavioral measures.

ELIGIBILITY:
Inclusion Criteria:

1. Ischemic or hemorrhagic stroke occurring at least 6 months prior to enrollment
2. Age range from 20 to 90 years
3. MMSE score < 28, or MoCA score < 25
4. Self- or informant-reported memory or cognitive complaints or Clinical dementia rating (CDR) scale ≤ 0.5
5. Able to follow the study instruction
6. Adequate cardiopulmonary function to perform aerobic exercise
7. Able to walk with or without assistive devices

Exclusion Criteria:

1. Unstable medical history (e.g., recent myocardial infarction) that might limit participation
2. Concomitant with other neurological disorders (e.g., Parkinson's disease, amyotrophic lateral sclerosis, multiple sclerosis)
3. Current participation in another interventional trial

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2018-08-30 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change scores of Mini-Mental State Exam (MMSE) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The Mini-Mental State Exam (MMSE) is used to screen patients for cognitive impairment, track changes in cognitive functioning over time, and often to assess the effects of therapeutic agents on cognitive function. Its range of total score is 0-30 with higher values indicating better cognitive function.
Change scores of the Montreal Cognitive Assessment (MoCA). | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The Montreal Cognitive Assessment (MoCA) will be used to assess general cognitive functions. It examines several cognitive domains with a total score of 30 and higher values indicate better cognitive functions. The MoCA has been shown to be a valid and promising tool to evaluate the global cognitive function in patients with stroke. The psychometric properties of MoCA are good to excellent for patients with cerebrovascular diseases.
Change scores of Wechsler Memory Scale - Third Edition (WMS-III) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  Several subtests of Wechsler Memory Scale - Third Edition (WMS-III) including Faces Recognition (total scale=48), Verbal Paired Associates (total scale = 32), Word Lists (total scale = 48), and Spatial Span (total scale=32) will be used to assess the immediate, delayed, and working memory tests. For each subtest, a higher number indicates better performance in memory function. The raw score of subtests will also be transferred to standardized Z scores and summed to represent an index of general memory function.
Change scores of Wechsler Adult Intelligence Scale - Third Edition (WAIS-III) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The Wechsler Adult Intelligence Scale - Third Edition (WAIS-III) is developed to measure an individual's intelligence level. The Digit Symbol-Coding (score range 0-133) and Matrix Reasoning (range 0-26) subtests will be used.A higher score indicating better performance. The raw score of each subtest will also be transferred to standardized Z scores and summed to represent an index of general cognitive function.
Change scores of Useful Field of View (UFOV) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The UFOV is a computer-based visual test containing three subtests: visuomotor processing speed, divided attention, and selective attention (Ball, Edwards, & Ross, 2007). The UFOV has been shown to have good test-retest reliability and validity to assess patients with stroke (George & Crotty, 2010).
Change scores of Stroop Color-Word Test | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The Stroop Color-Word test assesses the abilities of selective attention, inhibition and executive function. The participants will be tested under congruent and incongruent conditions. In the congruent condition, the participant will name the color ink of a word which is consistent with the written color name; whereas in the incongruent condition the participant will name the color ink differs from the written color name. In both conditions, the number of colors correctly named within 45 seconds will be measured and the performance in the congruent condition will be compared with the incongruent condition (Quaney et al., 2009).
Change scores of Dual-Task test | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The Dual-Task test evaluates the ability of set-shifting. Participants will sit and perform the box and block test (BBT) or walk 10 meters while doing secondary cognitive or motor tasks. Two cognitive secondary tasks will be performed by the participants: (1) arithmetic task: participants will be asked to perform serial subtractions by 7 starting from 100 or random two-digit numbers (e.g., Baetens et al., 2013); (2) tone discrimination task: participants will be presented a number of low and high-pitched tones and they will respond to either the high or low-pitched tones during the trial. Both cognitive task performances will be recorded and the results will be compared to single cognitive task performance. In addition to the cognitive dual-task, participants will perform a motor task (e.g., holding a cup of water) while walking.
Change scores of Timed Up and Go Test (TUG) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The TUG assesses the dynamic balance ability and mobility. The participants will be required to stand up from a chair, walk 3 meters, turn around, walk back to the chair, and sit down. The test-retest reliability of TUG on individuals with stroke was excellent (Ng & Hui-Chan, 2005).
Change scores of Six-Minute Walk Test (6MWT) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The 6MWT measures the maximum distance walked over 6 minutes, which assess the endurance and mobility level of the participants. The participants could rest as needed during the course of the test. The test-retest reliability and responsiveness has been established to be high for patients with chronic stroke (Fulk, Echternach, Nof, & O'Sullivan, 2008).
Change scores of Mobility Level | Baseline, posttest (an expected average of 3 months)
  Accelerometers will be used to provide an objective measure of the amount of arm movements in real-life situations. The participants will be asked to wear an Actigraphy activity monitor (ActiGraph, Shalimar, FL, USA) on both wrists for 3 consecutive days before and after training to measure the number of moves each minute, and the average counts of move per minute. The participants will be required to wear the device during the day except for doing water-based activities, such as bathing or swimming.The use of actigraphy to measure arm use and physical activity has been established for patients with stroke (Freedson, Melanson, & Sirard, 1998; Maguire et al., 2012).
Change scores of International Physical Activity Questionnaires (IPAQ) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The short form version of International Physical Activity Questionnaires (IPAQ) assesses sitting, walking, moderate-intensity activities and vigorous intensity activities. Frequency (measured in days per week) and duration (time per day) are collected separately and transferred to MET-minutes values for each specific type of activity. A combined total physical activity MET-min/week can be computed as the sum of Walking + Moderate + Vigorous MET-min/week scores. Higher total scores indicated more health-related activities.
Change scores of Fugl-Myer Assessment (FMA) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The upper limb subscale of the Fugl-Myer Assessment (FMA-UE) assesses the motor impairments of upper limbs after stroke. The FMA-UE contains 33 movements with a score range from 0 to 66. A higher score indicated better motor recovery in upper limbs.
Change scores of Rivermead Mobility Index (RMI) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The Rivermead Mobility Index (RMI) evaluates the participant's functional mobility, balance, gait and walking ability. It contains a 15-item scale which includes 14 questions and one direct observation, with a total of score of 15 and higher scores indicating better mobility performance.
Change scores of Muscle Strength | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  We will evaluate isometric knee flexors and extensors muscle strength using handheld dynamometer. Also, we will use hand dynamometer to measure grip strength of the affected and less affected hand while the participant is seated, with the elbow at 90-degree flexion. We will record the mean value of 3 attempts.
Change scores of Functional Independence Measure (FIM) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The FIM assesses the dependence level of individuals with stroke to perform 18 activities (13 motor and five cognitive tasks) in daily living. The score ranges from 18 to 126 and higher scores demonstrate greater independent participation in daily activities (Ottenbacher, Hsu, Granger, & Fiedler, 1996). The FIM has good interrater reliability and validity (Hsueh, Lin, Jeng, & Hsieh, 2002).
Change scores of Lawton Instrumental Activities of Daily Living Scale (Lawton IADL) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The Lawton IADL scale evaluates 8 activities with a score range from 0 to 8 (higher indicate better function). The inter-rater reliability and validity of the Lawton IADL have been established to be moderate to high for community-dwelling older adults (Graf, 2008; Lawton & Brody, 1969).
Change scores of Stroke Impact Scale (SIS) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The SIS contains 59 items measuring eight domains, including strength, hand function, ADL/IADL, mobility, communication, emotion, memory/thinking, and participation, with a single item assessing perceived overall recovery from stroke. The total score is the average of the domain scores, and the domain scores are the averages of the item scores (1-5), and higher scores indicate better function or QOL.
Change scores of EuroQol-5D Questionnaire (EQ-5D) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The quality of life will be assessed by the EQ-5D questionnaire which comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has three levels: no problems, some problems, extreme problems. The score has been shown to be reliable and valid (Greiner et al., 2003).
Change scores of Community Integration Questionnaire (CIQ) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The social participation level will be assessed with the Community Integration Questionnaire (CIQ).It contains 15 items to evaluate the degree of integration into each of the three area of family, social network, and productive activities. The total scores range from 0 to 29 with larger numbers indicating better integration.
Change scores of Geriatric Depression Scale (GDS) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The Geriatric Depression Scale (GDS) - 15 items version is a self-administered questionnaire used to evaluate mood and depressive symptoms. The scores range is 0-15 and a score of 5 or greater taken as a possible indicator of depression.
Task-based Electroencephalogram (EEG) | Baseline, posttest (an expected average of 3 months)
  The Task-based EEG will be collected when participants perform the n-back task before and after the intervention program to examine the effects of training on neural plasticity.
BDNF val66met genotype | Baseline
  Saliva samples will be collected at baseline to determine the Brain-Derived Neurotrophic Factor (BDNF) val66met genotype.
Serum BDNF level | Baseline, posttest (an expected average of 3 months)
  Blood samples will be collected at baseline and after the intervention programs. The blood tests will include serum BDNF level, antioxidative markers, HbA1C level, and Plasma lipid level.
  Serum BDNF will be quantified using an enzyme-linked immunosorbent assay (Human BDNF Quantitative Immunoassay, DBD00, R&D Systems) according to the manufacturer's instructions. This sandwich ELISA is set in order to measure natural and recombinant human mature BDNF in serum and plasma. All assays will be performed on F-bottom 96-well plates (Nunc, Wiesbaden, Germany).
Total antioxidant capacity (TAC) | Baseline, posttest (an expected average of 3 months)
  Blood samples will be collected at baseline and after the intervention programs. The blood tests will include BDNF level, antioxidative markers, HbA1C level, and Plasma lipid level.
  Antioxidative markers will be used to reflect the changes on oxidative stress. In particular, we will be analyzing the total antioxidant capacity (TAC).
Glucose indicator | Baseline, posttest (an expected average of 3 months)
  Blood samples will be collected at baseline and after the intervention programs. The blood tests will include BDNF level, antioxidative markers, HbA1C level, and Plasma lipid level.
  HbA1C level will be tested to investigate the relationships between blood glucose level and aerobic exercise.
Plasma lipid level | Baseline, posttest (an expected average of 3 months)
  Blood samples will be collected at baseline and after the intervention programs. The blood tests will include BDNF level, antioxidative markers, HbA1C level, and Plasma lipid level.
  The cholesterol ratio (total cholesterol divided by high-density lipid) will be evaluated to reflect the lipid level in the blood.

SECONDARY OUTCOMES:
Change scores of Caregiver Strain Index (CSI) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The Caregiver Strain Index (CSI) is a tool that can be used to quickly identify families with potential caregiving concerns. It is a 13-question tool that measures strain related to care provision. The reliability and validity has been established (Robinson, 1983).
Change scores of Caregiver Burden Scale(CBS) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  CBS evaluates the burden of the primary caregiver of the participants, including general strain, isolation, disappointment, emotional involvement, and environment of the caregivers. The CBS for caregivers of stroke patients showed moderate to good test-retest reliability and construct validity (Elmstahl, Malmberg, & Annerstedt, 1996).

CONTACTS AND LOCATIONS:
Overall Officials: Ching-yi Wu, ScD, Principal Investigator — Chang Gung Memorial Hospital
Locations (4):
- Taiwan (4):
  - Kaohsiung Municipal Siaogang Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Far Eastren Memorial Hospital, New Taipei City
  - Chang Gung Memorial Hospital, Taoyuan District